CLINICAL TRIAL: NCT02927847
Title: Targeting Reward Dysfunction as a Mechanism to Improve Smoking Cessation
Brief Title: Neuroimaging Reward, Behavioral Treatment, and Smoking Cessation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maggie M Sweitzer, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Maggie M Sweitzer, PhD, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00076408; K23DA039294 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BA + VLNC (Experimental): Participants will receive Nicotine Patch, SPECTRUM Nicotine Research Cigarettes (.03), and behavioral treatment prior to quit attempt, followed by standard nicotine replacement therapy with Nicotine Patch during the quit attempt. Behavioral treatments in this condition will include standard smoking cessation counseling plus behavioral activation therapy aimed at increasing reinforcement from non-drug rewards.
  Interventions: Drug: Nicotine Patch; Drug: SPECTRUM Nicotine Research Cigarettes (.03 mg); Behavioral: Behavioral Activation
- VLNC Only (Active Comparator): Participants will receive Nicotine Patch, SPECTRUM Nicotine Research Cigarettes (.03), and behavioral treatment prior to quit attempt, followed by standard nicotine replacement therapy with Nicotine Patch during quit attempt. Behavioral treatments in this condition will include standard smoking cessation counseling plus supportive counseling and health education.
  Interventions: Drug: Nicotine Patch; Drug: SPECTRUM Nicotine Research Cigarettes (.03 mg); Behavioral: Supportive Counseling

INTERVENTIONS:
Drug: Nicotine Patch — Both groups will receive nicotine patches (21 mg/d) to wear for 1 month prior to the quit date. After the quit date, both groups will wear the nicotine patch for 8 weeks (21 mg/d for 4 weeks, 14 mg/d for 2 weeks, and 7 mg/d for 2 weeks).
  Other Names: Nicoderm CQ
Drug: SPECTRUM Nicotine Research Cigarettes (.03 mg) — For 1 month prior to their quit date, participants will switch to smoking SPECTRUM Nicotine Research Cigarettes instead of their usual brand.
  Other Names: Very Low Nicotine Content Cigarettes
Behavioral: Behavioral Activation — Participants in the BA+VLNC group will undergo 8 60-minute behavioral sessions (4 pre-quit, 1 on quit day, and 3 post-quit) including 15 min of standard smoking cessation counseling and 45 minutes of behavioral activation treatment. BA components will include activity monitoring, values assessment, activity scheduling, and social contracts.
  Other Names: BA
  Arms: BA + VLNC
Behavioral: Supportive Counseling — Participants in the VLNC Only group will undergo 8 60-minute behavioral sessions (4 pre-quit, 1 on quit day, and 3 post-quit) including 15 min of standard smoking cessation counseling and 45 minutes of supportive counseling and health education. Supportive counseling and health education will include empathic listening as well as informational content on topics of exercise, nutrition, sleep and relaxation.
  Arms: VLNC Only

SUMMARY:
The goal of this study is to evaluate the effects of a smoking cessation intervention combining behavioral treatment with low nicotine cigarettes on neuroimaging measures of reward function and smoking cessation outcomes. The results of this study will provide information about mechanisms contributing to smoking and smoking cessation and will help to guide future treatment studies.

DETAILED DESCRIPTION:
Smokers who are interested in quitting will be randomly assigned to one of two treatment conditions. In the BA +VLNC condition (n = 16) smokers will switch to smoking very low nicotine cigarettes (VLNCs) while wearing a 21 mg/d nicotine patch for 5 weeks prior to their quit date. They will also participate in weekly behavioral activation (BA) treatment sessions. Smokers in the VLNC Only group (n = 19) will undergo the same pharmacological pretreatment but will undergo standard counseling and health education instead of BA. Following the quit date, both groups will receive standard nicotine replacement therapy. At baseline and pre-quit, BOLD response to smoking and non-smoking rewards will be measured using fMRI after 24 hr abstinence. Latency to relapse will serve as a continuous clinical outcome measure. Participants will also receive follow-up phone calls at 6 months and 12 months post-quit to assess smoking status.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* intact intellectual functioning (K-BIT2 >79)
* smoking at least 5 cigarettes per day
* expired CO concentration of at least 8 ppm or urinary cotinine > 100 ng/mL
* interested in quitting smoking

Exclusion Criteria:

* inability to attend all experimental sessions
* report of significant health problems
* use of psychoactive medications or current participation in psychotherapy
* current unstable psychiatric illness as assessed by clinical diagnostic interview
* suicidal ideation with plan or intent
* regular use of smokeless tobacco
* current alcohol or drug abuse
* use of illegal drugs (excluding marijuana) as measured by urine drug screen
* current use of nicotine replacement therapy or other smoking cessation treatment
* presence of contraindications for nicotine replacement therapy
* left-handed
* presence of conditions that would make MRI unsafe
* claustrophobia
* history of fainting
* pregnant, trying to become pregnant, or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2022-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggie M Sweitzer, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes): Participants will receive Nicotine Patch, SPECTRUM Nicotine Research Cigarettes (.03), and behavioral treatment prior to quit attempt, followed by standard nicotine replacement therapy with Nicotine Patch during the quit attempt. Behavioral treatments in this condition will include standard smoking cessation counseling plus behavioral activation therapy aimed at increasing reinforcement from non-drug rewards.
  Nicotine Patch: Both groups will receive nicotine patches (21 mg/d) to wear for 1 month prior to the quit date. After the quit date, both groups will wear the nicotine patch for 8 weeks (21 mg/d for 4 weeks, 14 mg/d for 2 weeks, and 7 mg/d for 2 weeks).
  SPECTRUM Nicotine Research Cigarettes (.03 mg): For 1 month prior to their quit date, participants will switch to smoking SPECTRUM Nicotine Research Cigarettes instead of their usual brand.
  Behavioral Activation: Participants in the BA+VLNC group will undergo 8 60-minute behavioral sessions (4 pre-quit, 1 on quit day, and 3 post-quit) including 15 min of standard smoking cessation counseling and 45 minutes of behavioral activation treatment. BA components will include activity monitoring, values assessment, activity scheduling, and social contracts.
- VLNC (Very Low Nicotine Cigarettes) Only: Participants will receive Nicotine Patch, SPECTRUM Nicotine Research Cigarettes (.03), and behavioral treatment prior to quit attempt, followed by standard nicotine replacement therapy with Nicotine Patch during quit attempt. Behavioral treatments in this condition will include standard smoking cessation counseling plus supportive counseling and health education.
  Nicotine Patch: Both groups will receive nicotine patches (21 mg/d) to wear for 1 month prior to the quit date. After the quit date, both groups will wear the nicotine patch for 8 weeks (21 mg/d for 4 weeks, 14 mg/d for 2 weeks, and 7 mg/d for 2 weeks).
  SPECTRUM Nicotine Research Cigarettes (.03 mg): For 1 month prior to their quit date, participants will switch to smoking SPECTRUM Nicotine Research Cigarettes instead of their usual brand.
  Supportive Counseling: Participants in the VLNC Only group will undergo 8 60-minute behavioral sessions (4 pre-quit, 1 on quit day, and 3 post-quit) including 15 min of standard smoking cessation counseling and 45 minutes of supportive counseling and health education. Supportive counseling and health education will include empathic listening as well as informational content on topics of exercise, nutrition, sleep and relaxation.
Period: Overall Study
Arm/Group | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) | VLNC (Very Low Nicotine Cigarettes) Only
Started | 16 | 19
Completed | 10 | 16
Not Completed | 6 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — PI withdrawn due to missed visits | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) | VLNC (Very Low Nicotine Cigarettes) Only | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (10.3) | 37.6 (8.5) | 37.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 14 | 16 | 30
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 9 | 13 | 22
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD (Blood-oxygen-level-dependent) Response to Monetary Reward
Description: Effects of BA+VLNC (vs. VLNC Only) on pre-quit changes in fMRI BOLD response to monetary reward anticipation. BOLD signal change is estimated from the contrast of monetary reward anticipation vs neutral anticipation, and extracted from voxels within the ventral striatum at each time point.
Time Frame: baseline, week 5
Population: Participants without good fMRI data at baseline or week 5 (due to missed session, signal dropout, or artifacts) are not included in analyses.
Measure: Mean (Standard Deviation); unit: fMRI BOLD signal
Arm/Group | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) | VLNC (Very Low Nicotine Cigarettes) Only
Number analyzed (Participants) | 10 | 14
fMRI BOLD signal | -0.085 (0.21) | -0.067 (0.36)
Statistical Analysis 1: Comparison: BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) vs VLNC (Very Low Nicotine Cigarettes) Only; Test type: Other; p = 0.891, t-test, 2 sided; t-value = 0.138

2. Primary Outcome: Change in BOLD (Blood-oxygen-level-dependent) Response to Smoking Reward
Description: Effects of BA+VLNC (vs. VLNC Only) on pre-quit changes in fMRI BOLD response to smoking reward anticipation. BOLD signal change is estimated from the contrast of smoking reward anticipation vs neutral anticipation, and extracted from voxels within the ventral striatum at each time point.
Time Frame: baseline, week 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fMRI BOLD signal
Arm/Group | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) | VLNC (Very Low Nicotine Cigarettes) Only
Number analyzed (Participants) | 10 | 14
fMRI BOLD signal | 0.011 (0.157) | -0.036 (0.226)
Statistical Analysis 1: Comparison: BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) vs VLNC (Very Low Nicotine Cigarettes) Only; Test type: Other; p = 0.571, t-test, 2 sided; t-value = -0.575

3. Primary Outcome: Number of Participants Who Relapsed or Are Presumed to Have Relapsed
Description: Relapse is defined as return to 7 consecutive days of smoking.
Time Frame: weeks 6 to 13
Measure: Count of Participants; unit: Participants
Arm/Group | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) | VLNC (Very Low Nicotine Cigarettes) Only
Number analyzed (Participants) | 16 | 19
Participants | 9 | 9
Statistical Analysis 1: Comparison: BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) vs VLNC (Very Low Nicotine Cigarettes) Only; Test type: Other; p = 0.739, Regression, Cox; Odds Ratio (OR) = 1.17

ADVERSE EVENTS:
Time Frame: Week 1 to week 13
Arm/Group | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) | VLNC (Very Low Nicotine Cigarettes) Only
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 13/16 | 16/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BA (Behavioral Activation) + VLNC (Very Low Nicotine Cigarettes) (N=16) | VLNC (Very Low Nicotine Cigarettes) Only (N=19)
Itchiness at patch site (Skin and subcutaneous tissue disorders) | 4 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Cold/upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Fever (Infections and infestations) | 0 | 1
Runny nose/congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Increased phlegm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Loss of voice (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mouth/throat irritaiton (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Heart burn (Gastrointestinal disorders) | 2 | 1
Hunger (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0
Stomach bug (Gastrointestinal disorders) | 3 | 1
Upset stomach/nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Headache (Nervous system disorders) | 3 | 3
Phantom Limb (Nervous system disorders) | 1 | 0
Heat sensitivity in extremeties (Nervous system disorders) | 1 | 0
Tightness in lower back (Musculoskeletal and connective tissue disorders) | 1 | 0
Hip pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthritis/joint pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Stress (Social circumstances) | 2 | 1
Vivid or abnormal dreams (General disorders) | 5 | 5
Insomnia (General disorders) | 2 | 3
Sleep issues (General disorders) | 1 | 0
Sedation (General disorders) | 0 | 1
Nicotine withdrawal (General disorders) | 1 | 0
Irritability (Psychiatric disorders) | 6 | 5
Jitteriness (Psychiatric disorders) | 1 | 0
Sadness (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Allergies/hay fever (Immune system disorders) | 1 | 2
Food allergy (Immune system disorders) | 1 | 0
Car accident (Injury, poisoning and procedural complications) | 1 | 0
Cut finger/hand (Injury, poisoning and procedural complications) | 0 | 2
Poison ivy (Injury, poisoning and procedural complications) | 1 | 0
Root canal (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and SAP (2018-08-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT02927847/Prot_SAP_000.pdf
  • Study Protocol: Study Protocol COVID Amendment (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT02927847/Prot_001.pdf